CLINICAL TRIAL: NCT03626870
Title: Effects of Resistin on Neutrophil Function
Status: Withdrawn | Type: Observational
Why Stopped: does not meet criteria for clinical trial
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Anthony Bonavia, Professor, Department of Anesthesiology, Penn State Health Milton S Hershey Medical Center
Other Study IDs: STUDY00010357
Record Dates: First submitted 2018-08-03; First posted 2018-08-13 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2023-03

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To assess the effect of resistin on neutrophil migration and intracellular bacterial killing

ELIGIBILITY:
Inclusion criteria:

* age ≥ 18
* gender: male or female

Exclusion Criteria

* Adults who are unable to provide informed consent themselves
* History of chronic kidney disease as defined by estimated glomerular filtration rate (GFR) <60 ml/min prior to cardiogenic shock
* Patients with hematologic malignancies
* Pregnant women
* Patient/surrogate is not fluent in English
* Long-term immunosuppressive therapy
* Prisoner
* Patients on pre-existing continuous reno-renal therapy (CRRT) or intermittent hemodialysis (IHD

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all healthy volunteer adults
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
intracellular bacterial killing, assessed by number of colonies of bacterial growth following neutrophil exposure to bacteria and resistin | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bonavia, MD, Principal Investigator — Penn State Milton S Hershey Med Ctr
Locations (1):
- Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No